CLINICAL TRIAL: NCT05516407
Title: A Phase I/II Open-Label Study to Evaluate the Safety and Efficacy of Orally Administered Full-Spectrum Medicinal Cannabis Plant Extract 0.08% THC (FEN164) in Children With Autism Spectrum Disorder.
Brief Title: Safety and Efficacy of Oral Full-Spectrum Medicinal Cannabis Plant Extract in Children With Autism Spectrum Disorder.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry); Monash Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNX001-21
Record Dates: First submitted 2022-04-04; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FEN164 (Experimental): Full-Spectrum Medicinal Cannabis Plant Extract with less than 0.08% THC (FEN164)
  Stage 1: 5mg/kg, 10mg/kg, 15mg/kg, 20mg/kg (1 week each) Stage 2: 20mg/kg (8 weeks), 15mg/kg, 10mg/kg, 5mg/kg (1 week each)
  Interventions: Drug: FEN164

INTERVENTIONS:
Drug: FEN164 — Oil based. Full-spectrum medicinal cannabis plant extract with less than 0.08% THC.

SUMMARY:
This is a 20-week open-label study to evaluate the safety and efficacy of full-spectrum medicinal cannabis plant extract < 0.08% THC (FEN164) in children with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
The study population will include twenty (20) boys and girls aged eight (8) years through to seventeen (17) years that have a medical diagnosis of Level 2 and 3 Autism Spectrum Disorder (ASD) as confirmed by the Autism Diagnostic Observational Schedule (ADOS-2) criteria.

Participants will commence treatment with a daily dose of 5mg/kg of FEN164. This will gradually increase over a four-week period until the maximum tolerated daily dose or 20mg/kg per day is achieved (Up-titration phase/Stage 1). Participants will continue to receive their respective maximum dose for eight (8) weeks (Treatment phase/Stage 2) which will be gradually decreased by 5 mg/kg for a period of 4 weeks until the end of the study (Down-titration phase).

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 8 years to 17 years (inclusive)
* Participant is at a healthy weight at the discretion of the Principal Investigator.
* Parents or caregivers can give informed consent for participation in the trial with assent from individuals with autism.
* Participants can comply with trial requirements.
* According the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria the participant has a diagnosis of Level 2 or 3 Autism Spectrum Disorder (ASD) confirmed by Autism Diagnostic Observational Schedule (ADOS-2) criteria
* All treatments including medications and therapies for ASD related symptoms must have been stable for 4 weeks before enrolment and for the duration of the trial wherever possible.
* Participants must be able to swallow liquid.
* Consent giver must be able to understand the requirements of the study.

Exclusion Criteria:

* Current diagnosis of bipolar disorder, psychosis, schizophrenia, schizoaffective disorder, or active major depression
* Has a diagnosis other than ASD that dominates the clinical presentation (e.g., Attention Deficit Hyperactivity Disorder [ADHD])
* Has a degenerative condition
* Changes in anticonvulsive therapy within the last 12 weeks
* Taking omeprazole, lansoprazole, tolbutamide, warfarin, sirolimus, everolimus, temsirolimus, tacrolimus, clobazam, repaglinide, pioglitazone, rosiglitazone, montelukast, bupropion, or efavirenz
* Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®, or Epidiolex®) within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients
* Participant has moderately impaired hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) or total bilirubin (TBL) > 2 × ULN. This criterion can only be confirmed once the laboratory results are available; participants enrolled into the trial who are later found to meet this criterion must be screen-failed.
* Participant is male and fertile (i.e., after puberty unless permanently sterile by bilateral orchidectomy) unless willing to ensure that they use male contraception (condom) or remain sexually abstinent during the trial and for 12 weeks thereafter.
* Participant is female and with childbearing potential (i.e., following menarche and until becoming postmenopausal for ≥ 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that they use a highly effective method of birth control (e.g., hormonal contraception, intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence) during the trial and for 12 weeks thereafter.
* Female participant who is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the trial or within 12 weeks thereafter.
* Participant had brain surgery or traumatic brain injury within 1 year of screening.
* Participant has any other significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.
* Any abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if they took part in the trial
* Any history of suicidal behaviour (lifelong) or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 4 weeks or at screening or randomization
* Participant has donated blood during the past 12 weeks and is unwilling to abstain from donation of blood during the trial.
* Participant has any known or suspected history of alcohol or substance abuse or positive drugs of abuse test at screening (not justified by a known concurrent medication).
* Participant has previously been enrolled into this trial.
* Participant has plans to travel outside their country of residence during the trial, unless the participant has confirmation that the product is permitted in the destination country/state

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale - Improvement (CGI-I) | Baseline, Weeks 5, 9, 13 & 17
  This is a 7-point scale measuring symptom change from baseline. Where a score of 1 is very much improved and a score of 7 is very much worse.

SECONDARY OUTCOMES:
Vineland Adaptive Behaviour Scales, Third Edition | Baseline, Week 17
  Used to measure adaptive functioning across three core domains (Communication, Daily Living Skills, and Socialization), and two optional domains (Motor Skills and Maladaptive Behaviour); items are rated on a 3-point scale (0=never; 1=sometimes; 2=usually or often). The core domains sum to a total Adaptive Behaviour Composite.
Social Responsiveness Scale, 2nd Editions (SRS-2) | Baseline, Week 17
  Five domains are assessed including: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behaviour. Items are scored on a 4-point scale (ranging from 1=not true to 4=almost always true).
Anxiety, Depression and Mood Scale (ADAMS) | Baseline, Week 17
  28 symptom items that resolve into five subscales labelled: Manic/Hyperactive Behaviour, Depressed Mood, Social Avoidance, General Anxiety, and Compulsive Behaviour. Items are rated on 4-point scale ranging from 0=not a problem to 3=severe problem.
Sleep Disturbance Scale for Children (SDSC) | Baseline, Weeks 5, 9, 13 & 17
  Six subscales including Disorders of Initiating and Maintaining Sleep, Sleep Breathing Disorders, Disorders of Arousal, Sleep Wake Transition Disorders, Disorders of Excessive Somnolence, and Sleep Hyperhydrosis. Items are rated on 5-point scale where 1=never and 5=always (daily). Subscale scores sum to equal a total score.
Clinical Global Impression-Severity (CGI-S) | Baseline, Weeks 5, 9, 13 & 17
  Reflects clinician's impression of severity of illness on a 7-point scale ranging from 1=not at all to 7=among the most extremely ill.
Autism Family Experience Questionnaire (AFEQ) | Baseline, Week 17
  Parent/Caregiver form used to measure impact of autism interventions on family experience and quality of life. Items are rated on a 5-point scale where 1=always and 5=never.
Anxiety Scale for Children - Autism Spectrum Disorder - Parent Version (ASC-ASD-P) | Baseline, Weeks 5, 9, 13 & 17
  Parent/Caregiver form developed to detect symptoms of anxiety in youth with ASD. Composed of four subscales (Performance Anxiety, Uncertainty, Anxious Arousal, and Separation Anxiety), items are rated on a 4-point scale (0=never and 3=always). Subscales sum to equal a total score.
Anxiety Scale for Children - Autism Spectrum Disorder - Child Version (ASC-ASD-C) | Baseline, Weeks 5, 9, 13 & 17
  Child form developed to detect symptoms of anxiety in youth with ASD. Composed of four subscales (Performance Anxiety, Uncertainty, Anxious Arousal, and Separation Anxiety), items are rated on a 4-point scale (0=never and 3=always). Subscales sum to equal a total score.
The Child Behaviour Checklist for Ages 6 - 18 (CBCL) | Baseline, Week 17
  A parent/carer measure to assess patterns of behaviour. The measure is a Likert scale rated over 3 or 4 points.
Caregiver Global Impression of Change in Attention (CGI-CA) | Baseline, Weeks 5, 9, 13 & 17
  Reflects clinician's impression of change in attention on a 7-point scale ranging from 1=not at all to 7=very severe problem. Provided as Baseline and Post-Baseline questionnaires.
Caregiver Global Impression of Change (CGI-C) Target Behaviour | Baseline, Weeks 5, 9, 13 & 17
  Reflects clinician's impression of change of behaviour on a 7-point scale ranging from 1=not at all to 7=very severe problem. Provided as Baseline and Post-Baseline questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fahey, Principal Investigator — Head of Paediatric Neurology
Locations (1):
- Monash Children's Hospital, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No